CLINICAL TRIAL: NCT06980948
Title: A Multicenter Phase 1 / 2 Double-blind, Randomized, Sham-controlled Dose Escalation Study to Determine Safety and Tolerability of Single Dose Intrathecal ST-503 Gene Therapy for Refractory Pain Due to Peripheral Neuropathy (Small Fiber Predominant, SFN)
Brief Title: Safety and Tolerability Study of ST-503 for Refractory Pain Due to Peripheral Neuropathy (Small Fiber Predominant, SFN)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-503-101
Record Dates: First submitted 2025-04-30; First posted 2025-05-20 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Chronic Neuropathic Pain
Keywords: Small Fiber Neuropathy
MeSH Terms: conditions — Small Fiber Neuropathy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, sham-controlled dose escalation study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Sham Controlled Study (Sham Comparator)
  Interventions: Procedure: Sham (No Treatment)
- Investigational Agent (Experimental)
  Interventions: Genetic: ST-503

INTERVENTIONS:
Genetic: ST-503 — Genomic Medicine
  Arms: Investigational Agent
Procedure: Sham (No Treatment) — Sham Procedure
  Arms: Sham Controlled Study

SUMMARY:
This research is being done to study a possible treatment for refractory pain due to small fiber neuropathy (SFN).

ST-503 is intended to deliver a modified copy of the gene which will ideally repress Nav1.7 tissue-related pain signals reaching the brain, which should reduce the refractory pain due to small fiber neuropathy (SFN).

DETAILED DESCRIPTION:
This research is being done to study a possible treatment for refractory pain due to small fiber neuropathy (SFN).

Small fiber neuropathy happens when something damages small nerve fibers in your skin, causing symptoms like painful tingling or burning sensations in your hands and feet. Pain originating in the nerves outside of the brain and spinal cord is defined by doctors as neuropathic pain. Scientists have discovered that certain proteins in our bodies called sodium channels are important for communicating pain signals in nerves, specifically, Nav1.7, Nav1.8 and Nav1.9.

This first-in-human study will test the use of a type of experimental treatment called "gene therapy." The primary goal is to determine if is safe and well tolerated. The second goal is to determine if it reduces the level of refractory pain due to SFN disease. The gene will be delivered into your cells using a special delivery tool called a vector.

ELIGIBILITY:
Inclusion Criteria

1. Signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
2. ≥ 18 years of age.
3. Diagnostic characterization of peripheral neuropathy (small fiber predominant) according to the Analgesic, Anesthetic, and Addiction Clinical Trial Translations, Innovations, Opportunities and Networks (ACTTION) criteria.

   a. Minimal large fiber polyneuropathy by clinical examination and by nerve conduction studies (NCS) during screening. NCS results may be based on unilateral assessment. However, bilateral SNAP responses must be within normal range for age and gender in the ulnar, radial, and sural nerves to enhance sensitivity of monitoring for DRG ganglionopathy post ST-503 dosing or sham procedure treatment. Only persons with normal SNAP responses may be enrolled.
4. An IENFD punch skin biopsy demonstrating reduction below the 5th percentile of sex and age-adjusted normal values must be performed and sent for IENFD evaluation at the Cutaneous Nerve Lab at University of Utah.
5. Medical record documentation that pain is refractory to 2 of 3 categories of first line medical therapy for at ≥ 6 months prior to screening.

   a. "Refractory to first line medical therapy" is defined as failure to have an average weekly pain score < 5 after an adequate trial of two of three categories of first line medication treatments for neuropathic pain (tricyclic antidepressants, SNRI, or gabapentinoids).
6. Average PI-NRS score ≥ 5 over seven-day pain assessment interval.

   1. Minimum acceptable PI-NRS reporting requirement for eligibility: Four of seven days with two daily PI-NRS scores (morning and afternoon) must be recorded with a single PI-NRS score (morning or afternoon) for the remaining three days.
   2. Subjects will not be told at any time that the eligibility requirement is an average PI-NRS ≥ 5, to avoid biasing the pain intensity scoring during the screening and baseline periods.
7. Body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 40 kg/m2
8. Agreement to limit alcohol consumption to not more than one 12 oz beer, 5 oz glass of wine, or 2 oz of liquor daily for a minimum of two months after the procedure.
9. Negative screening test for mycobacterium tuberculosis (MTB) within 1 year prior to consent.
10. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria

1. Serum sample positive for pre-existing anti-AAV9 antibodies per predefined cut point based on assay sensitivity.
2. Drug- and alcohol-related:

   1. Persons using opioid analgesics for under 3 months or persons who are not on a stable dose of opioids; if on a stable dose, the dose may decrease over the course of the study but should not be increased.
   2. History of known alcohol abuse, opioid analgesic abuse, or illicit drug abuse within 2 years of Screening.
   3. Positive urine test for drugs of abuse (including opiates, benzodiazepines, amphetamines, cocaine, barbiturates, and phencyclidine) without prescription and investigator approval, at Screening and Day -1.
   4. Use of cannabinoids is not permitted.
3. Persons with Fabry disease, fibromyalgia, peripheral neuropathies due to alcohol or drug toxicity, or diagnosed channelopathies (congenital insensitivity to pain, inherited erythromelalgia).
4. Corticosteroid-related:

   1. Use of glucocorticoids except for topical or ophthalmic preparations within 6 weeks prior to screening visit
   2. Hypersensitivity or contraindications to corticosteroid use including but not limited to clinically significant osteoporosis, uncontrolled hypertension, poorly controlled diabetes, uncontrolled hyperlipidemia, or hypercholesterolemia
5. Neurologic-related:

   1. Subjects with severe pain conditions other than SFN which would interfere with clinical study assessments
   2. Documented stroke or transient ischemic attack within 1 year prior to consent
   3. History of poorly controlled epilepsy or recurrent unexplained blackouts
6. Procedure-related:

   1. Contraindications to LP, general anesthesia or sedation
   2. Any medical disorders that, in the opinion of the Investigator, could interfere with LP including but not limited to evidence for a pressure gradient between supratentorial and infratentorial compartments, Arnold-Chiari malformation, bleeding diathesis, clinically significant coagulopathy, thrombocytopenia, increased intracranial pressure, or spine disease or past surgical procedures involving the spine
7. Infectious disease-related:

   a. Active viral infection or bacterial infection including but not limited to the following:

   i. Active Hepatitis A, B, or C infection
   * Patients with previous, adequately resolved hepatitis A, B or C are eligible for the study
   * Patients with chronic hepatitis B or C are not eligible for the study

     b. A severe infection (e.g., pneumonia, septicemia, central nervous system infections [e.g., meningitis, encephalitis]) within 12 weeks prior to Screening

     c. Patients who receive COVID-19 vaccine or booster will have a waiting period of 4 weeks or more before they may be dosed with ST-503, so that the vaccine response does not interfere with the gene therapy and vice versa. They should not receive a COVID-19 vaccine or booster within 4 weeks after subjects have been dosed with ST-503. Subjects should not receive any live-attenuated vaccine, for any disease, 2 weeks before and 20 weeks after the ST-503 or sham procedure administration.
8. Endocrine-related:

   a. History or evidence of impaired glucose metabolism based on hemoglobin A1C level of ≥ 6.5%
9. Cardiac- and circulatory system-related:

   1. History of unstable angina, myocardial infarction, or chronic heart failure within 1 year prior to consent
   2. Clinically significant primary valvular heart disease and/or prosthetic cardiac valve
   3. 12-lead ECG demonstrating QTcF (Fridericia's correction) > 450 msec

   i. If QTcF exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTcF values should be used to determine the subject's eligibility. The ECG can be repeated after the subject is supine for 10 minutes. A third ECG can be obtained after an additional 10 minutes while remaining supine.

   d. Presence of uncontrolled hypertension
10. Hepatic disease- and hepatotoxic medication-related:

    1. Presence of clinically relevant liver disease
    2. Hepatic dysfunction as indicated by one or more of the following:

    i. Albumin ≤ 3.5 g/dL ii. Total bilirubin > 1.5 x ULN and direct bilirubin ≥ 0.5 mg/dL iii. ALP > 2 x ULN iv. ALT or AST > 1.5 x ULN

    c. Hepatotoxic medications should be avoided during the study period including acetaminophen exceeding 4 gm/day unless essential to patient's treatment, approved by investigator, and hepatic dysfunction is not identified

    d. Hepatotoxic supplement use during the study period
11. Hematologic-related:

    1. Personal or family history of coagulopathy
    2. Presence of condition or treatment associated with increased bleeding risk associated with LP
    3. Hematocrit < 35% (assigned male at birth) or < 32% (assigned female at birth)
    4. Absolute neutrophil count < 2000 cells/µL
    5. International normalized rate (INR) above normal range for lab at study site
    6. Platelet count below laboratory lower limits of normal (LLN)
12. Renal-related:

    a. History of chronic renal disease or creatinine ≥ 1.5 mg/dL
13. Cancer-related:

    a. History of cancer, including B-cell cancers, within 5 years of Screening i. Exceptions to this exclusion are fully excised non-melanoma skin cancers, non-metastatic prostate cancer, and fully treated ductal carcinoma in situ of the breast, provided subject has been stable for at least 6 months
14. Allergy- and immunology-related:

    1. History of severe allergic or anaphylactic reactions
    2. History of hypersensitivity to any inactive ingredient of the IP or to corticosteroids
    3. Chronic autoimmune disease that is being treated with immunosuppressants, including but not limited to corticosteroids
    4. Previous autologous or allogeneic bone marrow transplant, peripheral stem cell transplant or solid organ transplantation
15. Previously received gene or cellular therapy
16. Participation in other interventional studies during the period of current study participation
17. Planned surgery within three months prior to consent or during the study
18. Any active legal action related to pain disorder
19. Any other reason that, in the opinion of the Site Investigator or the Study Medical Monitor, would render the subject unsuitable for participation in the study. A suicide risk of imminent risk of self-harm according to the C-SSRS is an exclusion criterion for the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) | 12 weeks
  To assess safety and tolerability of ST-503 over a 12-week post-dosing observation period.

SECONDARY OUTCOMES:
Percentage of subjects with pain intensity reduction from baseline at Week 12 | 12 weeks
  * 30% in the weekly average of daily pain intensity measurements performed using the PI-NRS
  * 50% in the weekly average of daily pain intensity measurements performed using the PI-NRS
    * Dose of rescue medication use
    * Frequency of rescue medication use
Percentage of subjects at Week 12 | 12 weeks
  * Categorized as improved on the patient global impression of change (PGIC) assessment
  * With a ≥ 1-point improvement in suicidal ideation in Columbia Suicide Severity Rating Scale (C-SSRS) responses
Columbia Suicide Severity Rating Scale (CSSRS) Rating | 12 weeks
  With a ≥ 1-point decline in suicidal ideation in Columbia Suicide Severity Rating Scale (CSSRS) responses
Overall Pain Intensity Numerical Rating Scale (PI-NRS) score | 12 Weeks
  Participants will rate their pain intensity using an 11-point Numerical Rating Scale (0=no pain and 10=worst possible pain) and record their score in an electronic diary.
Short Form McGill Pain Questionnaire-2 (SF-MQ-2) | 12 Weeks
  This pain scale was developed to evaluate chronic neuropathic and non-neuropathic pain in adults. It consists of 22 descriptors of pain in 4 parts (continuous, intermittent, neuropathic, and affective pain types) to be rated from 0-10 with 0 indicating no pain and 10 the worst pain ever during the past week.
Daily Sleep Interference Score (DSIS) | 12 Weeks
  DSIS is assessed on an 11-point NRS, which ranges from 0 (none) to 10 (severe).
Hospital Anxiety and Depression Scale (HADS) | 12 Weeks
  HADS is a screening tool for anxiety and depression in non-psychiatric clinical populations consisting of 14 items (seven each for anxiety and depression). Higher scores correlate with worse symptoms.
Rasch-Transformed 13-item SFN Symptoms Inventory Questionnaire | 12 Weeks
  The 13-item SFN-SIQ evaluates changes in physiological functions such as sweating patterns and incontinence using a four-point Likert scale (0 = never present, 1 = sometimes, 2 = often, and 3 = always present) to get a sum of the grading scores attributed to each of the 13 items with a 0 to 39 range. Higher scores correlate with worse symptoms.
SFN-specific Rasch-built Overall Disability Scale (SFN-RODS) | 12 Weeks
  The 32-item SFN-RODS is a disease-specific interval measure suitable to detect activity limitations and participation restrictions in patients with SFN. The scale ranges from 0 to 64 with higher numbers indicating worse disability.
36-Item Short Form Health Survey (SF-36) domains and summary scores | 12 Weeks
  This measures quality of life measures such as physical functioning, emotional well-being, energy levels, and social functioning. The range is from 0-100 with higher scores being associated with a better perceived quality of life.
Pain Catastrophizing Questionnaire (PCS) | 12 Weeks
  PCS has 13 questions related to rumination, magnification and helplessness with values ranging 0 to 4 for a total possible score of 52. The higher the score the more pain catastrophizing is present.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics Inc.
Locations (10):
- United States (10):
  - HonorHealth, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No